CLINICAL TRIAL: NCT06555809
Title: Pharmacokinetic Evaluation of Artesunate in Infants Being Treated for Severe Malaria - Research Laboratory Addendum to the Observational Study Titled: Safety and Efficacy of Artesunate in Pregnant Women and Infants (< One Month of Age)
Brief Title: Evaluation of Artesunate in Infants Being Treated for Severe Malaria
Status: Recruiting | Type: Observational
Sponsor: Amivas Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IVAS-PEDS-PK-1
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Malaria
Keywords: Artesunate; Infant
MeSH Terms: conditions — Malaria | interventions — Artesunate; Injections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Artesunate Injection — Additional blood sample will be collected when other standard of care blood specimens are collected during the 2-day period after the start of intravenous artesunate treatment.
  Other Names: Artesunate for Injection

SUMMARY:
This is essentially a laboratory study that is an addendum to an ongoing prospective Phase 4 multicenter observational study titled: "Safety and Efficacy of Artesunate in Pregnant Women and Infants (ARTEMUM)" being conducted in France. Infants, the parents of whom provided consent to have data collected from their child as part of the ARTEMUM study, will have an additional blood sample collected when other standard of care blood specimens are collected during the 2-day period after the start of intravenous (IV) artesunate treatment. A maximum of 4 samples will be taken and plasma will be isolated and stored frozen until analysis for plasma artesunate and dihydroartemisinin (DHA) concentrations. Red blood cells will also be frozen for further analysis (for example Kelch-13 mutations). In addition, a standard of care blood sample will be collected approximately one month post treatment for clinical laboratory tests.

DETAILED DESCRIPTION:
This is essentially a laboratory study that is an addendum to an ongoing prospective Phase 4 multicenter observational study titled: "Safety and Efficacy of Artesunate in Pregnant Women and Infants (ARTEMUM)" being conducted in France. Parents of infants under 2 years of age who provided consent to participate in the ARTEMUM study will be asked to provide consent for their child to this laboratory study providing the infant was eligible for the ARTEMUM study. During the first 48 hours after the start of IV artesunate treatment, a maximum of 4 samples of blood will be collected when other standard of care samples are being collected. With regard to blood collected for standard of care, it is recognized that samples between 0.25 and 5 hours post doses will be the most useful for pharmacokinetic (PK) analysis due to the 30-to-45-minute half-life of DHA. Plasma will be isolated and frozen until submission to the central laboratory for artesunate and DHA plasma concentrations. In addition, a standard of care blood sample will be collected approximately one month post treatment for clinical laboratory tests. The recommendation by the World Health Organization (WHO) is followed in France not only for safety (anemia) but also for relapse. Clinical laboratory test results and other data to be included in the analysis will be abstracted from the case report forms (CRFs) from the ARTEMUM study.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent provided to the ARTEMUM Study
* Parental consent provided to participate in this PK Laboratory Study
* Infants < 2 years of age with malaria (positive blood by polymerase chain reaction (PCR) or thin or thick smear or rapid diagnostic test (RDT), or any combination of those) treated by at least 1 dose of intravenous artesunate

Exclusion Criteria:

* Hemoglobin < 7.0 g/dL at the time when additional blood sample for PK assessment will be drawn as part of standard of care

Ages: 1 Minute to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants < 2 years of age with malaria (positive blood by PCR or thin or thick smear or RDT treated with at least 1 dose of intravenous artesunate with hemoglobin (Hb) levels ≥ 7.0 g/dL.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-10-06 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in concentration of artesunate in blood plasma samples | Approximately at 5 minutes, 30 minutes, 90 minutes, and 4 hours after artesunate intravenous injection
  Change in concentration of artesunate in blood plasma samples collected as part of standard of care
Change in concentration of dihydroartemisinin in blood plasma samples | Approximately at 5 minutes, 30 minutes, 90 minutes, and 4 hours after artesunate intravenous injection
  Change in concentration of dihydroartemisinin in blood plasma samples collected as part of standard of care

SECONDARY OUTCOMES:
Safety, as measured by the number of participants with adverse events | During standard of care treatment with intravenous artesunate
  Safety, as measured by the number of participants with adverse events
Tolerability, as measured by the number of doses of artesunate administered to each participant | During standard of care treatment with intravenous artesunate
  Tolerability of artesunate treatment, as measured by the number of doses of artesunate administered to each participant

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Smith, MD, Principal Investigator — Amivas Inc.
Locations (1):
- Hôpital Cochin Port Royal, Paris, France

IPD SHARING:
Plan to Share IPD: No